CLINICAL TRIAL: NCT06029244
Title: Eyecontrol coMmunication Platform for dEliRium manaGemEnt in Intensive Care Units (EMERGE) : A Multicenter Randomized Controlled Trial
Brief Title: Eyecontrol coMmunication Platform for dEliRium manaGemEnt in Intensive Care Units (EMERGE)
Acronym: EMERGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: BIRD (Israel-United States Binational Industrial Research and Development) Foundation- Funding agency (Unknown); Rabin Medical Center (Other); Assuta Medical Center (Other); Eyefree Assisting Communication Ltd (Industry)
Responsible Party: Principal Investigator, Somnath Bose, MD, Assistant Professor of Anesthesia, Harvard Medical School, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023P000563
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Delirium; Delirium in Old Age; Critical Illness; Intensive Care Unit Delirium
MeSH Terms: conditions — Delirium; Critical Illness

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to either a) EyeControl-Pro assisted active intervention arm or b) sham control
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be unblinded, or unmasked, to treatment allocation given the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EyeControl-Pro assisted active intervention arm (Active Comparator): Participants will wear the EyeControl-Pro device daily from 08:00-18:00 (extendable to 20:00; minimum 4 hours for compliance). On Day 1, onboarding includes a ≤2 min auditory tutorial, repeated daily for orientation. The device delivers up to 5 personalized family messages and 5 automated re-orientation messages per day, alternating approximately every 2 hours to maintain engagement and awareness. Slow-tempo music or white/brown noise plays in 15-minute sessions every 4 hours, modulated according to the patient's preferences and responses. The device performs twice-daily automated CAM-ICU assessments, scheduled within 45 minutes of blinded assessor CAM-ICU to allow comparison. Study team delirium assessments occur twice daily through Day 7, then once daily if in ICU for days 8-14, with MoCA/t-MoCA and HADS at Day 30 (+14 day window). Device use ends after 7 days, earlier if extubated, discharged, transitioned to comfort care, or in the event of death.
  Interventions: Device: EyeControl-Pro
- Sham Control (Sham Comparator): Participants will wear an identical-appearing EyeControl device daily from 08:00-18:00 (extendable to 20:00; minimum 4 hours for compliance). On Day 1, onboarding includes a ≤2 min auditory tutorial introducing the device. No automated re-orientation messages, family messages, or music sessions are delivered. The device tracks eye state and logs activity but does not provide auditory feedback beyond the initial tutorial. Blinded study team members perform twice-daily CAM-ICU and CAM-ICU-7 assessments through Day 7, then once daily if in ICU for days 8-14. MoCA/t-MoCA and HADS assessments occur at Day 30 (+14 day window). Device is removed after 7 days, upon extubation, ICU discharge, comfort care transition, or death.
  Interventions: Other: Control

INTERVENTIONS:
Device: EyeControl-Pro — Based on artificial intelligence (AI)-powered eye-tracking technology, the EyeControl-Pro wearable device and smart platform enable 24/7 customizable communication and monitoring between ventilated patients who cannot speak, their families, and medical teams
  Arms: EyeControl-Pro assisted active intervention arm
Other: Control — No intervention
  Arms: Sham Control

SUMMARY:
The purpose of this research is to investigate whether addition of the EyeControl-Pro platform as an adjunct to standard guideline-based intensive care unit management of critically ill patients is effective in reducing delirium incidence and severity.

DETAILED DESCRIPTION:
This is a prospective, binational, single-blind, multicenter, randomized control trial, conducted according to international good clinical practice (GCP) ethical and quality standards. Critically ill, mechanically ventilated patients aged >=50 years with Richmond Agitation Sedation Scale (RASS) score of -3 to +1 (at time of screening) who are anticipated to require ventilation for >=24 hours will be eligible for recruitment. The study will be conducted simultaneously at Beth Israel Deaconess Medical Center (BIDMC) Boston, USA, Assuta Ashdod Medical Center (Ashdod, Israel) and Rabin Medical Center (Petah Tikvah, Israel) with BIDMC contributing up to 50% of the total enrollment. Participants will be randomized to either a) sham device or b) active intervention arm (details described below). Legally appointed representatives, patients and caregiver teams will be administered an optional questionnaire to assess their experience with the study device at the conclusion of the study protocol. Study subjects will be administered the telephone-Montreal Cognitive Assessment (t-MoCA); total score of 22 - missing 8 points present in Montreal Cognitive Assessment (MoCA) pertaining to drawing/executive function not feasible over phone) or MoCA (if still in-hospital; assessed out of total score of 30) and Hospital Anxiety and Depression Scale (HADS) questionnaire 30 days post-randomization. Hebrew versions of these questionnaires will be used at Israeli sites.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients aged >=50 years
* RASS score of -3 to +1 and
* Anticipated to require >=24 hours of mechanical ventilation

Exclusion Criteria:

* Not expected to survive >=24 hours
* Have limitations in care (Do Not Resuscitate, or comfort-focused care orders)
* Receiving paralytic neuromuscular blocking agent (NMBA) infusion or anticipated need for NMBA use
* Have advanced dementia or cognitive impairment including post-concussive syndrome.
* Have severe uncorrected psychiatric disorders.
* Have uncorrected hearing or visual impairment.
* Acute or subacute neurological disorder hindering communication or ability to participate in CAM ICU assessments
* Enrolled in a clinical trial which prohibits co-enrollment.
* Incarcerated
* Have no identified legally appointed representative (LAR)
* Are unable to communicate in the predominant local language (English at US site and English/Hebrew/Arabic/Russian in Israel)
* Refusal of treating clinical team.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of any delirium occurrence defined as CAM ICU 7 score (>=2) during the first 7 days in ICU post-randomization or ICU discharge/death (whichever is sooner) | Upto 7 days or liberation from ventilator whichever is sooner.
  To evaluate if study subjects randomized to active EyeControl-Pro arm have a higher proportion of delirium free assessments as assessed by CAM (confusion assessment method)-ICU 7 during device usage for up to 7 days when compared with those in the sham EyeControl-Pro arm. CAM-ICU is a validated assessment tool for detection of ICU delirium.

SECONDARY OUTCOMES:
Prevalence of severe delirium assessments (defined as CAM ICU 7>=6) during the first 7 days in ICU post-randomization or ICU discharge/death (whichever is sooner) | Upto 7 days or discharge from intensive care unit (ICU) whichever is sooner
  To evaluate if study subjects in the active EyeControl-Pro arm have lower prevalence of severe delirium assessments as measured by CAM-ICU7 within first 7 days post randomization or ICU discharge (whichever is sooner) when compared to sham control arm. CAM-ICU 7 is a validated instrument for measurement of delirium severity with scores ranging from 0-7.
Mean number of days with delirium (defined as the total number of days with at least one CAM ICU 7 positive delirium assessment within 7 days post-randomization or up to discharge from the ICU/death, whatever occurs earlier. | Upto 7 days or discharge from intensive care unit (ICU) whichever is sooner
  To evaluate if subjects randomized to the active EyeControl-Pro arm have lower delirium incidence (as measured by CAM-ICU) within first 7 days post randomization or ICU discharge whichever is sooner when compared to sham EyeControl-Pro arm.

OTHER OUTCOMES:
Cognitive scores | 30 days post-randomization.
  To compare cognitive function at 30 days post enrollment using the t-MoCA (telephone-Montreal Cognitive Assessment) or MoCA (if still in-hospital) questionnaire. MoCA is a validated instrument for assessment of cognition with range 0-30 (0-22 for telephonic version) score of over 26 indicates normal.
Depression anxiety scores | 30 days post-randomization.
  To compare depression and anxiety scores at 30 days post enrollment using the HADS (Hospital Anxiety and Depression Scale) questionnaire.HADS ranges from 0-21 with higher scores indicating worse depression or anxiety
CAM ICU concordance | During device usage upto 7 days
  Agreement between CAM ICU assessment between Eyecontrol and investigator administered CAM-ICU in active intervention arm
Days free of restraints | Upto 7 days or discharge from intensive care unit
  Comparison of days free of restraints between 2 groups
Use of rescue medications for delirium and agitation | Upto 7 days or discharge from intensive care unit
  Use of medications for agitated delirium
ICU days alive and free of delirium and coma | Upto 7 days or discharge from intensive care unit (ICU) whichever is sooner
  To evaluate if subjects randomized to the active EyeControl-Pro arm have higher number of days free of coma and delirium within first 7 days post randomization or ICU discharge whichever is sooner when compared to sham EyeControl-Pro arm

CONTACTS AND LOCATIONS:
Overall Officials: Somnath Bose, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States
- Israel (2):
  - Assuta Ashdod Medical Center, Ashdod
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Girard TD, Pandharipande PP, Ely EW. Delirium in the intensive care unit. Crit Care. 2008;12 Suppl 3(Suppl 3):S3. doi: 10.1186/cc6149. Epub 2008 May 14. PMID 18495054
- [Background] Mart MF, Williams Roberson S, Salas B, Pandharipande PP, Ely EW. Prevention and Management of Delirium in the Intensive Care Unit. Semin Respir Crit Care Med. 2021 Feb;42(1):112-126. doi: 10.1055/s-0040-1710572. Epub 2020 Aug 3. PMID 32746469
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Smith CD, Grami P. Feasibility and Effectiveness of a Delirium Prevention Bundle in Critically Ill Patients. Am J Crit Care. 2016 Dec;26(1):19-27. doi: 10.4037/ajcc2017374. PMID 27965224
- [Background] Kinchin I, Mitchell E, Agar M, Trepel D. The economic cost of delirium: A systematic review and quality assessment. Alzheimers Dement. 2021 Jun;17(6):1026-1041. doi: 10.1002/alz.12262. Epub 2021 Jan 21. PMID 33480183
- [Background] Hayhurst CJ, Pandharipande PP, Hughes CG. Intensive Care Unit Delirium: A Review of Diagnosis, Prevention, and Treatment. Anesthesiology. 2016 Dec;125(6):1229-1241. doi: 10.1097/ALN.0000000000001378. PMID 27748656
- [Background] Pun BT, Badenes R, Heras La Calle G, Orun OM, Chen W, Raman R, Simpson BK, Wilson-Linville S, Hinojal Olmedillo B, Vallejo de la Cueva A, van der Jagt M, Navarro Casado R, Leal Sanz P, Orhun G, Ferrer Gomez C, Nunez Vazquez K, Pineiro Otero P, Taccone FS, Gallego Curto E, Caricato A, Woien H, Lacave G, O'Neal HR Jr, Peterson SJ, Brummel NE, Girard TD, Ely EW, Pandharipande PP; COVID-19 Intensive Care International Study Group. Prevalence and risk factors for delirium in critically ill patients with COVID-19 (COVID-D): a multicentre cohort study. Lancet Respir Med. 2021 Mar;9(3):239-250. doi: 10.1016/S2213-2600(20)30552-X. Epub 2021 Jan 8. PMID 33428871
- [Background] Nikooie R, Neufeld KJ, Oh ES, Wilson LM, Zhang A, Robinson KA, Needham DM. Antipsychotics for Treating Delirium in Hospitalized Adults: A Systematic Review. Ann Intern Med. 2019 Oct 1;171(7):485-495. doi: 10.7326/M19-1860. Epub 2019 Sep 3. PMID 31476770
- [Background] Neufeld KJ, Yue J, Robinson TN, Inouye SK, Needham DM. Antipsychotic Medication for Prevention and Treatment of Delirium in Hospitalized Adults: A Systematic Review and Meta-Analysis. J Am Geriatr Soc. 2016 Apr;64(4):705-14. doi: 10.1111/jgs.14076. Epub 2016 Mar 23. PMID 27004732